CLINICAL TRIAL: NCT03865576
Title: Validation of a Non-Invasive Intracranial Pressure (ICP) Device by Comparison With Implanted Intracranial Pressure Monitoring Instrumentation or Lumbar Puncture
Brief Title: Validation of Non-Invasive Intracranial Pressure (ICP) Monitoring Device
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston Neurosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: nICP-1
Record Dates: First submitted 2019-02-28; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Intracranial Hypertension; Abnormality of Intracranial Pressure
Keywords: ICP; Papilledema; Neurological Intensive Care
MeSH Terms: conditions — Intracranial Hypertension; Papilledema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Thomas Jefferson University: Patients in intensive care with altered intracranial pressure.
  Intervention: Non-invasive ICP measurement using transorbital Doppler ultrasound device.
  Comparison of measurements obtained with values derived from surgically implanted ICP monitoring sensors.
  Interventions: Diagnostic Test: Non-invasive ICP measurement
- Honor Health in Phoenix: Patients in intensive care with altered intracranial pressure.
  Intervention: Non-invasive ICP measurement using transorbital Doppler ultrasound device.
  Comparison of measurements obtained with values derived from surgically implanted ICP monitoring sensors.
  Interventions: Diagnostic Test: Non-invasive ICP measurement
- Emory University Hospital in Atlanta: Patients in intensive care with altered intracranial pressure.
  Intervention: Non-invasive ICP measurement using transorbital Doppler ultrasound device.
  Comparison of measurements obtained with values derived from surgically implanted ICP monitoring sensors
  Interventions: Diagnostic Test: Non-invasive ICP measurement
- University of Washington: Patients in intensive care with altered intracranial pressure.
  Intervention: Non-invasive ICP measurement using transorbital Doppler ultrasound device. .
  Comparison of measurements obtained with values derived from surgically implanted ICP monitoring sensors and lumbar puncture
  Interventions: Diagnostic Test: Non-invasive ICP measurement

INTERVENTIONS:
Diagnostic Test: Non-invasive ICP measurement — Intracranial pressure will be measured non-invasively using transorbital Doppler ultrasound. Values will be compared to ICP measured by lumbar puncture or implanted ICP sensors

SUMMARY:
For purposes of validation, this study compares intracranial pressure measurements obtained with a novel self-calibrating, non-invasive, intracranial pressure measuring (ICP) device, with the values obtained from (a) patients in an intensive care unit (ICU) whose meet standard clinical indications for ICP measurement and whose ICP is measured using gold-standard implanted intracranial instrumentation and in (b) ambulatory subjects who meet clinical indications for lumbar puncture.

DETAILED DESCRIPTION:
This study is designed to validate intracranial pressure measurements obtained with a novel, self-calibrating, non-invasive, intracranial pressure measuring (ICP) device based on trans-cranial Doppler technology. The ophthalmic artery is utilized as a natural ICP sensor. Up to 80 subjects will be recruited in 4 centers to achieve a power of 90% and a p<0.05 compared to the values obtained from (a) patients in an ICU whose meet standard clinical indications for ICP measurement and whose ICP is measured using gold-standard implanted intracranial instrumentation and in (b) ambulatory subjects who meet clinical indications for lumbar puncture. At least two comparative readings, separated by an hour or more, will be obtained from each subject.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients suspected of having an abnormality of ICP undergoing monitoring with commercially-available, FDA-approved instrumentation.

Exclusion Criteria:

History of:

* Glaucoma or optic hypertension
* Severe orbital or ophthalmic injury
* Orbital or intraocular surgery that might interfere with orbital compliance
* Congenital malformations of the eye and/or orbit that might interfere with orbital compliance or orbital vascular anatomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in an ICU who meet clinical criteria for invasive ICP measurement,
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Non-invasive intracranial pressure (ICP) value | Up to 5 days after admission to ICU
  ICP value measured using novel non-invasive measurement device
Second non-invasive intracranial pressure (ICP) value | Up to 6 days after admission to ICU
  A second measurement of ICP using novel non-invasive ICP measurement device

CONTACTS AND LOCATIONS:
Overall Officials: T Forcht Dagi, MD, DMedSc, Study Director — Boston Neurosciences
Locations (4):
- United States (4):
  - Honor Health Research Institute, Phoenix, Arizona
  - Emory University Hospital, Atlanta, Georgia
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No